CLINICAL TRIAL: NCT04333771
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Clinical Study to Evaluate the Efficacy and Safety of SHR0302 in Moderate to Severe Active Rheumatoid Arthritis Subjects With Inadequate Response to csDMARDs.
Brief Title: A Study to Evaluate the Efficacy and Safety of SHR0302 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR0302-301
Record Dates: First submitted 2020-04-02; First posted 2020-04-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- SHR0302 dose1 (Experimental)
  Interventions: Drug: SHR0302
- SHR0302 dose2 (Experimental)
  Interventions: Drug: SHR0302

INTERVENTIONS:
Drug: SHR0302 — The placebo group will take drugs orally for 24 weeks, and then switch to SHR0302 dose1 for 28 weeks, in the meanwhile, SHR0302 dose1 group and SHR0302 dose2 group will continue taking drugs for the whole 52 weeks.
  Arms: SHR0302 dose1; SHR0302 dose2
Drug: Placebo — The placebo group will take drugs orally for 24 weeks, and then switch to SHR0302 dose1 for 28 weeks, in the meanwhile, SHR0302 dose1 group and SHR0302 dose2 group will continue taking drugs for the whole 52 weeks.
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy and safety of different doses of JAK1 inhibitor SHR0302 in subjects with moderate to severe active rheumatoid arthritis who had inadequate response to conventional synthetic DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent.
* RA diagnosis consistent with the 2010 ACR/EULAR criteria;
* Moderate to severe RA defined by 6 or more tender joints, 6 or more swollen joints (68- or 66-joint count), and an ESR of 28 mm/h or greater or a CRP level greater than 5mg/L.
* Subjects were required to have an inadequate response to treatment with csDMARDs before baseline.
* If subjects are taking permitted csDMARDs or low-dose corticosteroid orally at baseline , the stable doses should have lasted for more than 4 weeks already.
* BMI ≥18 kg/m2

Exclusion Criteria:

* Pregnant women or refuse to receive contraception during the study.
* Lab abnormality within 4 weeks of randomization as follows: WBC count <3.0×10^9/L；neutrophil count<1.5×10^9/L;hemoglobin level<90.0 g/L ; platelet count <100×10^9/L; AST or ALT levels greater than the upper limit of normal; HBsAg or HCV or HIV antibody positivity.
* History of another autoimmune rheumatic disease ; history of cancer or infection including tuberculosis and hepatitis; history of important cardiovascular events or thrombotic diseases.
* Previous treatment with JAK inhibitor or cytotoxic drugs; bDMARDs within 6 months of randomization; other strong immunosuppressants within 3 months of randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
ACR20 response rate at week 24 | Week 24
  Response rate of 20% improvement in American College of Rheumatology (ACR20) criteria at week 24

SECONDARY OUTCOMES:
ACR20 response rate at week 52 | Week 52
  Response rate of 20% improvement in American College of Rheumatology (ACR20) criteria at week 52
ACR50 response rate at week 24 and week 52 | Week 24 and week 52
  Response rate of 50% improvement in American College of Rheumatology (ACR50) criteria at week 24 and week 52
ACR70 response rate at week 24 and week 52 | Week 24 and week 52
  Response rate of 70% improvement in American College of Rheumatology (ACR70) criteria at week 24 and week 52
Change from baseline in HAQ-DI score at week 24 and week 52 | Week 24 and week 52
  Change from baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) score at week 24 and week 52
Change from baseline in SF-36 score at week 24 and week 52 | Week 24 and week 52
  Change from baseline in the medical outcomes study 36-Item Short-Form Health Survey (SF-36) score at week 24 and week 52
DAS28-CRP <2.6 proportion at week 24 and week 52 | Week 24 and week 52
  Disease Activity Score for 28-joint counts based on the c-reaction protein (DAS28-CRP) of less than 2.6
DAS28-CRP≤3.2 proportion at week 24 and week 52 | Week 24 and week 52
  Disease Activity Score for 28-joint counts based on the c-reaction protein (DAS28-CRP) of equal to and less than 3.2

CONTACTS AND LOCATIONS:
Locations (1):
- Liuzhou workers' Hospital, Liuchow, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu J, Jiang Y, Zhang S, Liu S, Su J, Lin C, He X, Wu R, Yang L, Liu H, Duan X, Xu S, Luo H, Liu J, Xie Q, Mi C, Chen L, Zhang N, Gong H, Zhu J, Li Y, Wei H, Qian L, Wang J, Shi X, Jin H, Jiang Z, Xie X, Zhan F, Geng X, Zheng Z, Du Z, Dong G, Sun Y, Zeng X. Ivarmacitinib, a selective Janus kinase 1 inhibitor, in patients with moderate-to-severe active rheumatoid arthritis and inadequate response to conventional synthetic DMARDs: results from a phase III randomised clinical trial. Ann Rheum Dis. 2025 Feb;84(2):188-200. doi: 10.1136/ard-2024-226385. Epub 2025 Jan 3. PMID 39919893